CLINICAL TRIAL: NCT05860062
Title: Evaluation of Vitamin D Supplementation in Patients With Episodic and Chronic Tension-type Headache.
Brief Title: Vitamin D Supplementation in Episodic and Chronic Tension-type Headache
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Especialidades, Centro Medico Nacional "La Raza", Instituto Mexicano del Seguro Social (Other)
Responsible Party: Principal Investigator, Mario Mireles, Head of the Division of health research, Hospital de Especialidades, Centro Medico Nacional "La Raza", Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-2023-1301-045
Record Dates: First submitted 2023-04-24; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Chronic Tension-Type Headache
MeSH Terms: interventions — Vitamin D; Cholecalciferol; Calcium

STUDY DESIGN:
Intervention Model Description: The patients selected as the study population will be randomly distributed using a random number table, giving them the number 1, 2 or 3, according to the treatment group they will belong to.
Who Masked: Participant, Investigator
Masking Description: Each month the treatment will be given in equal bottles that will be marked on the label with a color (red, blue, green), the green color corresponding to placebo, red to vitamin D3+calcium and blue to calcium, only the doctors in charge of applying the questionnaires will know the group to which each patient belongs, in this way the double blind is not broken.
  The placebo will be used to evaluate the effect that produced the feeling of being benefited from a new treatment, the foregoing to avoid bias and have greater reliability of the results, when compared with the gold standard.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- calcium+topiramate/amitriptyline (Placebo Comparator): Patients with prophylactic treatment (amitriptyline, topiramate) + and Calcium: 1 Tablet every 24 hours containing: Calcium Carbonate 300 mg + Calcium Lactate Gluconate 2.94 g (500 mg of calcium).
  Interventions: Other: Calcium
- vitamin D3/calcium+topiramate/amitriptyline, (Experimental): Patients with prophylactic treatment (amitriptyline, topiramate) + Vitamin D and calcium supplementation: 1 Tablet every 24 hours containing: Calcium carbonate 1666.670 mg (600 mg calcium) + Vitamin D3 6.2 mg (400 IU).
  Interventions: Dietary Supplement: Vitamin D; Other: Calcium
- vitamin D+topiramate/amitriptyline (Active Comparator): Patients with prophylactic treatment (amitriptyline, topiramate) + 0.266 mg of calcifediol (15,960 IU of vitamin D)
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — Patients with prophylactic treatment (amitriptyline, topiramate) + 0.266 mg of calcifediol (15,960 IU of vitamin D)
  Other Names: colecalciferol
  Arms: vitamin D+topiramate/amitriptyline; vitamin D3/calcium+topiramate/amitriptyline,
Other: Calcium — 3: Patients with prophylactic treatment (amitriptyline, topiramate) + and Calcium: 1 Tablet every 24 hours containing: Calcium Carbonate 300 mg + Calcium Lactate Gluconate 2.94 g (500 mg of calcium).
  Arms: calcium+topiramate/amitriptyline; vitamin D3/calcium+topiramate/amitriptyline,

SUMMARY:
The goal of this clinical trial is to learn about the effect of vitamin D in patients with prophylactic therapy for episodic and chronic tension-type headache in amitriptyline or topiramate treatment. The main question it aims to answer are:

• What is the effect of vitamin D in patients with prophylactic therapy for episodic and chronic tension-type headache?

Patients will have the next selection criteria:

* Patients diagnosed by a neurologist in the headache clinic
* Criteria for episodic and chronic tension-type headache
* Poor clinical response to prophylactic treatment (amitriptyline, topiramate)
* Use of at least 1 prophylactic medication or a history of having used them.
* Onset of disease between the ages of 18 and 60
* Signature of informed consent

The population will be randomly divided into the following 3 treatment groups:

* Participants amitriptyline or topiramate treatment.
* Patients with placebo (Calcium) + topiramate/amitriptyline,
* Participants with vitamin D3/calcium+topiramate/amitriptyline. Researchers will compare the groups to see if vitamin D can decrease the intensity of your headache and therefore have a new therapeutic option.

DETAILED DESCRIPTION:
It will be a 4 month study. Each month a package containing treatment will be delivered, which may be conventional medication or tablets with conventional medication added with vitamins.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed by a neurologist in the headache clinic
* Criteria for episodic and chronic tension-type headache
* Poor clinical response to prophylactic treatment (amitriptyline, topiramate)
* Use of at least 1 prophylactic medication or a history of having used them.
* Onset of disease between the ages of 18 and 60
* Signature of informed consent

Exclusion Criteria:

* Patients with secondary headache (cranioencephalic trauma, cerebral infarction)
* Patients with primary headache other than tension headache
* Suffer heart, liver, and kidney diseases.
* Medications: thiazides
* Pregnant women
* They do not want to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2023-09-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Headache Impact Test, HIT-6 | 4 months
  It consists of 6 questions, assesses the frequency and severity of headaches in general in the last month. Emphasizes the frequency of severe forms of each headache, if it prevents you from doing homework, work or school, if you need to lie down, tiredness, irritability or difficulty concentrating in the last month. The answers will be quantified in: Never (0 points), almost never (5 points), sometimes (10 points), frequently (15 points), always (20 points) and the points of the 6 questions were added. With a total of 48 points or less, it is determined according to the questionnaire that there is no functional limitation, with points between 50 and 60 it is advisable to go to a doctor, between 50 and 54 the impact of disability is slight, from 55 to 68 the impact is moderate and over 60 the impact is severe.

SECONDARY OUTCOMES:
Depression Beck's Depression II | 4 months
  It is a self-report composed of 21 Likert-type items, used to detect and assess the severity of depression. Each item is answered on a 4-point scale, from 0 to 3, except for items 16 (changes in sleep pattern) and 18 (changes in appetite) which contain 7 categories. If a person chooses several response categories in an item, the category that corresponds to the highest score will be taken. At the end, the points of the 21 items will be added. The minimum and maximum scores on the test are 0 and 63.
  Cut-off points have been established that allow those evaluated to be classified into one of the following four groups: 0-13, minimal depression; 14-19, mild depression; 20-28, moderate depression; and 29-63, severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Jose J García, Dr., Study Director — Hospital de Especialidades
Locations (1):
- Hospital de Especialidades, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No